CLINICAL TRIAL: NCT02981628
Title: A Phase 2 Study of Inotuzumab Ozogamicin (NSC# 772518) in Children and Young Adults With Relapsed or Refractory CD22+ B-Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Inotuzumab Ozogamicin in Treating Younger Patients With B-Lymphoblastic Lymphoma or Relapsed or Refractory CD22 Positive B Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AALL1621; NCI-2016-01494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AALL1621 (Other: Children's Oncology Group); AALL1621 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia; Recurrent B Lymphoblastic Lymphoma; Refractory B Acute Lymphoblastic Leukemia; Refractory B Lymphoblastic Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — asparaginase erwinia chrysanthemi recombinant; Asparaginase; Specimen Handling; Biopsy; calaspargase pegol; Cyclophosphamide; Cytarabine; X-Rays; Inotuzumab Ozogamicin; Leucovorin; Spinal Puncture; Methotrexate; merphos; pegaspargase; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (inotuzumab ozogamicin) (Experimental): Patients receive inotuzumab ozogamicin IV over 60 minutes on days 1, 8, and 15 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. (COMPLETE)
  Interventions: Biological: Inotuzumab Ozogamicin
- Cohort II (inotuzumab ozogamicin, mBFM chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Asparaginase Erwinia chrysanthemi; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration and Biopsy; Drug: Calaspargase Pegol; Drug: Cyclophosphamide; Drug: Cytarabine; Procedure: Diagnostic Imaging Testing; Biological: Inotuzumab Ozogamicin; Drug: Leucovorin Calcium; Procedure: Lumbar Puncture; Drug: Methotrexate; Drug: Pegaspargase; Drug: Vincristine

INTERVENTIONS:
Drug: Asparaginase Erwinia chrysanthemi — Given Asparaginase Erwinia chrysanthemi
  Other Names: Asparaginase Erwinia chrysanthemi (Recombinant)-rywn; Asparaginase Erwinia chrysanthemi, Recombinant-rywn; Asparaginase Erwinia chrysanthemi-rywn; Crisantaspase; Crisantaspase Biobetter JZP-458; Crisantaspasum; Enrylaze; Erwinase; Erwinaze; JZP 458; JZP-458; JZP458; PF743; RC-P JZP-458; Recombinant Asparaginase erwinia chrysanthemi JZP-458; Recombinant Crisantaspase JZP-458; Recombinant Erwinia asparaginase JZP-458; Rylaze
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Procedure: Bone Marrow Aspiration and Biopsy — Undergo a bone marrow aspiration and biopsy
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Drug: Calaspargase Pegol — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol-mknl; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Drug: Cytarabine — Given IV or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Procedure: Diagnostic Imaging Testing — Undergo imaging
  Other Names: Diagnostic Imaging; Medical Imaging
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC 544; CMC-544; CMC544; Way 207294; WAY-207294
Drug: Leucovorin Calcium — Given PO or IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Drug: Pegaspargase — Given IV or IM
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)
Drug: Vincristine — Given IV
  Other Names: LCR; Leurocristine; VCR; Vincrystine
  Arms: Cohort II (inotuzumab ozogamicin, mBFM chemotherapy)

SUMMARY:
This phase II trial studies how well inotuzumab ozogamicin works in treating younger patients with B-lymphoblastic lymphoma or CD22 positive B acute lymphoblastic leukemia that has come back (relapsed) or does not respond to treatment (refractory). Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a toxic agent called ozogamicin. Inotuzumab attaches to CD22 positive cancer cells in a targeted way and delivers ozogamicin to kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the morphologic response rate (complete response [CR] + complete response with incomplete hematologic recovery [CRi]) following one cycle of treatment with inotuzumab ozogamicin in children with relapsed or refractory CD22+ B acute lymphoblastic leukemia (B-ALL). (Cohort 1)

SECONDARY OBJECTIVES:

I. To determine the CR/CRi rate following 2 cycles of inotuzumab ozogamicin therapy. (Cohort 1) II. To determine the safety of single agent inotuzumab ozogamicin administered at the adult recommended phase 2 dose (RP2D) to pediatric patients with relapsed or refractory CD22+ B-ALL. (Cohort 1) III. To determine the level of minimal residual disease (MRD) by flow cytometry in responding patients. (Cohorts 1 and 2) IV. To determine the incidence, severity, and outcomes of sinusoidal obstruction syndrome (SOS) of the liver in patients during inotuzumab ozogamicin therapy and following subsequent treatment, including myeloablative hematopoietic stem cell transplantation (HSCT). (Cohorts 1 and 2) V. To estimate the 3-year event-free survival (EFS), 3-year overall survival (OS), and among responders, duration of CR/CRi for pediatric patients with relapsed or refractory B-ALL treated with inotuzumab ozogamicin. (Cohort 1) VI. To describe inotuzumab ozogamicin pharmacokinetics and immunogenicity in pediatric patients in the presence of overt leukemia and in remission. (Cohort 1) VII. To determine the safe and tolerable dose of inotuzumab ozogamicin in combination with the augmented modified Berlin-Frankfurt-Munster (mBFM) consolidation chemotherapy backbone. (Cohort 2)

EXPLORATORY OBJECTIVES:

I. To describe the levels of leukemic blast CD22 surface expression and site density, and to explore the correlation with cytogenetics and clinical outcomes after treatment with inotuzumab ozogamicin. (Cohorts 1 and 2) II. To explore potential mechanisms of resistance to inotuzumab ozogamicin therapy including CD22 splice variants and intracellular signaling pathways. (Cohorts 1 and 2) III. To explore the impact of inotuzumab ozogamicin on humoral immune function and peripheral B cell populations. (Cohorts 1 and 2) IV. To describe the level of MRD by next-generation high-throughput sequencing (HTS) techniques which may detect low level leukemic blast populations that have altered CD22 expression. (Cohorts 1 and 2) V. To prospectively explore candidate SOS biomarkers including the endothelial marker of inflammation Angiopoietin 2 (Ang2) and the hepatic specific complement marker L-ficolin. (Cohorts 1 and 2) VI. To explore the use of prophylactic ursodeoxycholic acid (UDCA) to prevent hepatic damage and SOS during inotuzumab ozogamicin therapy and subsequent HSCT. (Cohorts 1 and 2) VII. To describe the interaction between inotuzumab ozogamicin and chimeric antigen receptor (CAR) T cell therapy before or after treatment with inotuzumab ozogamicin. (Cohorts 1 and 2) VIII. To estimate the CR/CRi rate following one cycle of inotuzumab ozogamicin plus augmented mBFM consolidation chemotherapy (first 42 days) and following 2 cycles within the confines of a pilot study. (Cohort 2)

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive inotuzumab ozogamicin intravenously (IV) over 60 minutes on days 1, 8, and 15 of each cycle. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. (COMPLETE)

COHORT II: Patients receive inotuzumab ozogamicin IV over 60 minutes on days 1, and 8. Patients also receive cyclophosphamide IV over 30-60 on day 1; cytarabine IV over 1-30 minutes or subcutaneously (SC) on days 1-4 and 8-11; leucovorin calcium orally (PO) or IV on days 2, 9, 16, 23 and 37 of cycle 1 and days 9 and 37 of cycle 2; pegaspargase or calaspargase pegol IV over 1-2 hours or pegaspargase intramuscularly (IM) on day 15; and vincristine IV on days 15 and 22. Patients receive methotrexate intrathecally (IT) on days 1, 8 and 36 of cycle 1 and day 36 of cycle 2 for CNS 1 patients, days 1, 8, 15, 22 and 36 of cycle 1, and day 36 of cycle 2 for CNS 2 patients. CNS 3 patients receive methotrexate intrathecal triple therapy (ITT) IT on days 1, 8, 15, 22 and 36 of cycle 1 and days 8 and 36 of cycle 2. There are 3 dose levels. If excessive toxicity is observed at dose level 1, the dosing of inotuzumab ozogamicin will be decreased for dose level -1 and 6-mercaptopurine omitted. If excessive toxicity is observed at this dose, then for dose level -2, the dosing of inotuzumab ozogamicin and cyclophosphamide will be decreased. Treatment repeats every 42 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow aspiration or biopsy, lumbar puncture, and blood sample collection throughout the trial. Patients also undergo imaging on screening and on study.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 1 year, and then yearly for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 1 year and < 22 years of age at the time of enrollment
* Patients must have B-ALL, or previously diagnosed B lymphoblastic lymphoma (B-LL), with >= 5% (M2 or M3) bone marrow blasts with or without extramedullary disease

  * NOTE: Relapsed patients previously diagnosed with B-lymphoblastic lymphoma (B-LL) are eligible if they have an M2 or M3 marrow at the time of enrollment on this study
* Patients with ALL or B-LL who have M2 morphology must have local confirmatory testing showing >= 5% blasts by flow cytometry, fluorescence in situ hybridization (FISH) testing or other molecular method
* Leukemic blasts must demonstrate surface expression of CD22 at the time of relapse by local/institutional flow cytometry of a bone marrow aspirate sample; (assessment of CD22 using a bright fluorophore such as phycoerythrin [PE] is strongly recommended)

  * In the case of an inadequate aspirate sample (dry tap) or if bone marrow aspirate is unable to be performed due to patient clinical status, flow cytometry of peripheral blood specimen may be substituted if the patient has at least 1,000/uL circulating blasts; alternatively, CD22 expression may be documented by immunohistochemistry of a bone marrow biopsy specimen
* Patients with one of the following:

  * Second or greater relapse;
  * Primary refractory disease with at least 2 prior induction attempts;
  * First relapse refractory to at least one prior re-induction attempt
  * Any relapse after HSCT (Cohort 1 ONLY)

Patients with Down syndrome are eligible ONLY for Cohort 1 with:

* Any of above disease status, OR
* First relapse with no prior re-induction attempt NOTE: Patients with Down syndrome or prior HSCT are NOT eligible for Cohort 2 combination therapy

  * Patients with Philadelphia chromosome (Ph)+ ALL must have had two prior therapy attempts including two different tyrosine kinase inhibitors (TKIs)
  * Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy, defined as resolution of all such toxicities to =< grade 2 or lower per the inclusion/exclusion criteria prior to entering this study. Apply to Cohort 2:
* Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned Research Coordinator prior to enrollment.

  * A waiting period prior to enrollment is not required for patients receiving standard cytotoxic maintenance chemotherapy (i.e., corticosteroid, vincristine, 6MP, and/or methotrexate).
  * A waiting period is not required for patients receiving a single dose of intrathecal methotrexate, hydrocortisone, and/or cytarabine within 7 days prior to enrollment
  * >= 14 days must have elapsed after the completion of other cytotoxic therapy, with the exception of hydroxyurea, for patients not receiving standard maintenance therapy. For patients who previously received calaspargase pegol, >= 21 days must have elapsed after the last dose. Additionally, patients must have fully recovered from all acute toxic effects of prior therapy.

    * Note: Cytoreduction with hydroxyurea must be discontinued >= 24 hours prior to the start of protocol therapy.
* Anti-cancer agents not known to be myelosuppressive (e.g., not associated with reduced platelet or absolute neutrophil count [ANC] counts): >= 7 days after the last dose of agent. For agents not listed, the duration of this interval must be discussed with the study chair and the study-assigned research coordinator prior to enrollment.
* Anti-cancer agents that are antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1. There is an exception for blinatumomab infusions, for which patients must have been off for at least 3 days and all drug related toxicity must have resolved to grade 2 or lower as outlined in the inclusion/exclusion criteria.
* Corticosteroids: If used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid. A waiting period prior to enrollment is not required for patients receiving corticosteroid for leukemia therapy/cytoreduction.
* Radiotherapy: >= 2 weeks must have elapsed since local palliative radiation therapy (XRT) (small port); >= 3 months must have elapsed if prior cranial or craniospinal XRT was received, if >= 50% of the pelvis was irradiated, or if total body irradiation (TBI) was received; >= 6 weeks must have elapsed if other substantial bone marrow irradiation was given.
* Stem cell transplant or rescue without TBI: For Cohort 1, at least 90 days must have elapsed since stem cell transplant and at least 30 days from donor lymphocyte infusion. Patient must have had no more than one previous HSCT and currently have no evidence of active graft vs. host disease (GVHD). For Cohort 2, no prior HSCT is allowed.
* Chimeric antigen receptor (CAR) T cell therapy: At least 30 days must have elapsed from the last CAR-T cell infusion

  * Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
  * Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or
  * A serum creatinine based on age/gender as follows:
* 1 to < 2 years: maximum serum creatinine 0.6 mg/dL (both male and female)
* 2 to < 6 years: maximum serum creatinine 0.8 mg/dL (both male and female)
* 6 to < 10 years: maximum serum creatinine 1 mg/dL (both male and female)
* 10 to < 13 years: maximum serum creatinine 1.2 mg/dL (both male and female)
* 13 to < 16 years: maximum serum creatinine 1.5 mg/dL (male), 1.4 mg/dL (female)
* >= 16 years: maximum serum creatinine 1.7 mg/dL (male), 1.4 mg/dL (female)

  * Direct bilirubin =< 1.5 x upper limit of normal (ULN) for age, and
  * Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 5 x ULN for age; for the purpose of this study, the ULN for ALT will be 45 U/L

Exclusion Criteria:

* Patients with any prior history of SOS irrespective of severity
* Patients with isolated central nervous system (CNS), testicular, or any other extramedullary site of relapse
* Patients who have been previously treated with inotuzumab ozogamicin
* Patients who have previously received HSCT (Cohort 2 only)
* Patients with Down syndrome (Cohort 2 only)
* History of allergic reaction attributed to compounds of similar or biologic composition to inotuzumab ozogamicin or other agents in the study

  * Note: Patients with history of allergy to pegaspargase/calaspargase pegol are eligible for enrollment on Cohort 2 if Erwinia formulation of asparaginase can be obtained
* Patients with active optic nerve and/or retinal involvement are not eligible; patients who are presenting with visual disturbances should have an ophthalmologic exam and, if indicated, a magnetic resonance imaging (MRI) to assess optic nerve or retinal involvement
* Patients who are currently receiving another investigational drug
* Patients who are currently receiving or plan to receive other anti-cancer agents (except hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy, and intrathecal chemotherapy)
* Anti-GVHD or agents to prevent organ rejection post-transplant; patients who are receiving cyclosporine, tacrolimus, or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant are not eligible for this trial; at least 3 half-lives must have elapsed after the last dose of GVHD or anti-rejection medications
* Patients who are currently receiving or plan to receive corticosteroids except as described below

  * Systemic corticosteroids may be administered for cytoreduction up to 24 hours prior to the start of protocol therapy, (Cohort 1 only) for all patients, corticosteroids may be administered as a premedication for inotuzumab ozogamicin and as treatment for allergic reactions or for physiologic replacement/stress dosing of hydrocortisone for documented adrenal insufficiency; corticosteroids are not allowed for other indications
* Patients with known human immunodeficiency virus (HIV), hepatitis B or C infections; testing to prove negative status is not required for enrollment unless it is deemed necessary for usual medical care of the patient
* Patients who have an active uncontrolled infection defined as:

  * Positive bacterial blood culture within 48 hours of study enrollment;
  * Fever above 38.2 degree Celsius (C) within 48 hours of study enrollment with clinical signs of infection; fever that is determined to be due to tumor burden is allowed if patients have documented negative blood cultures for at least 48 hours prior to enrollment and no concurrent signs or symptoms of active infection or hemodynamic instability
  * A positive fungal culture within 30 days of study enrollment or active therapy for presumed invasive fungal infection
  * Patients may be receiving IV or oral antibiotics to complete a course of therapy for a prior documented infection as long as cultures have been negative for at least 48 hours and signs or symptoms of active infection have resolved; for patients with clostridium (C.) difficile diarrhea, at least 72 hours of antibacterial therapy must have elapsed and stools must have normalized to baseline
  * Active viral or protozoal infection requiring IV treatment
* Patients known to have one of the following concomitant genetic syndromes: Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Schwachman (Schwachman-Diamond-Blackfan) syndrome or any other known bone marrow failure syndrome
* There have been no human studies of inotuzumab ozogamicin in pregnant women and no reports of exposure in utero; based on nonclinical safety studies, inotuzumab ozogamicin has the potential to impair human male and female fertility and to adversely affect human embryo fetal development; women of childbearing potential should be advised to avoid becoming pregnant while receiving inotuzumab ozogamicin; there is no information regarding the presence of inotuzumab ozogamicin in human milk, the effects on the breast-fed infant, or the effects on milk production; because of the potential for adverse reactions in breast-fed infants, women should not breast-feed during treatment with inotuzumab ozogamicin and for at least 2 months after the final dose

  * Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained within 7 days prior to enrollment
  * Female patients who are sexually active and of reproductive potential are not eligible unless they agree to use an effective contraceptive method for the duration of their study participation and for 8 months after the last dose of inotuzumab ozogamicin
  * Men with female partners of childbearing potential should use effective contraception during treatment with inotuzumab ozogamicin and for at least 5 months after the last dose of inotuzumab ozogamicin
  * Lactating females are not eligible unless they agree not to breastfeed their infants

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Morphologic response (complete response [CR]+ incomplete hematologic recovery [CRi]) following one cycle of treatment with inotuzumab ozogamicin (Cohort 1) | Up to 28 days
  The response rate will be estimated using the proportion of eligible/evaluable patients with CR/CRi response. A one-sided lower 95% Agresti-Coull confidence limit will be calculated.

SECONDARY OUTCOMES:
Morphologic response (CR + CRi) following 2 cycles of inotuzumab ozogamicin therapy (Cohort1) | Up to 56 days
  The response rate will be estimated using the proportion of eligible/evaluable patients with CR/CRi response.
Incidence of dose-limiting toxicities at recommended phase II dose (RP2D) (Cohort 1) | During Cycle 1, up to 28 days
  Evaluated according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicity tables will be constructed to summarize the observed incidence by type of toxicity and grade. For a given reporting period, a patient will be counted only once for a given toxicity for the worst grade of that toxicity reported for that patient.
Level of minimal residual disease (MRD) assessed in bone marrow by flow cytometry (Cohort 1 and 2) | Up to 2 cycles
  MRD negativity rates (< 0.01% detectable leukemia cells) will be estimated.
Incidence of adverse events of sinusoidal obstruction syndrome (SOS) of liver (Cohort 1 and 2) | Up to 1 year from last dose of Inotuzumab ozogamicin
  Evaluated according to NCI CTCAE version 5.0. The incidence of SOS of the liver in patients during inotuzumab ozogamicin therapy and following subsequent treatment including myeloablative hematopoietic cell transplantation (HSCT) will be described.
Event free survival (EFS) (Cohort 1) | From study entry to first event (induction failure, induction death, relapse, second malignancy, remission death), or date of last follow-up for event free subjects, assessed up to 3 years
  The EFS rate will be estimated using Kaplan Meier approach.
Overall survival (OS) (Cohort 1) | From the time from study entry to death or date of last follow-up, assessed up to 3 years
  The OS rate will be estimated using Kaplan Meier approach.
Duration of CR, CRi (Cohort 1) | Up to 3 years
  Among responding patients, three-year complete continuous response will also be estimated using duration of CR/CRi for the overall responding group and stratified by whether or not the patients proceed to HSCT.
Pharmacokinetic (PK) parameters, i.e., inotuzumab ozogamicin trough levels (Cohort 1) | Cycles 1 and 2 (each cycle is 28 days)
  Inotuzumab ozogamicin trough levels (ng/mL) will be determined in serum by validated, high sensitivity liquid chromatography-mass spectrometry (LCMS) assays. Descriptive summary statistics will be provided for the trough levels at scheduled visits for Cycles 1 and 2.
Immunogenicity (Cohort 1) | Cycles 1 and 2
  Enhanced chemiluminescence (ECL) and cell-based assays will be used to detect anti-drug antibodies and neutralizing antibodies to inotuzumab ozogamicin in serum. Inotuzumab ozogamicin trough levels will be compared between patients with and without antibodies.
Incidence of dose-limiting toxicities at the selected dose level of inotuzumab ozogamicin in combination with the augmented modified Berlin-Frankfurt-Munster (mBFM) consolidation chemotherapy (Cohort 2) | Up to cycle 1 (each cycle is 42 days)
  Evaluated according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicity tables will be constructed to summarize the observed incidence by type of toxicity and grade. For a given reporting period, a patient will be counted only once for a given toxicity for the worst grade of that toxicity reported for that patient.

OTHER OUTCOMES:
Changes in CD22 surface expression (Cohorts 1 and 2) | Baseline, post Cycle 1, and at time of relapse
  Exploratory analysis of CD22 will focus primarily on the comparison of paired pre-treatment and post-treatment samples at the following times, 1) End of cycle 1 and 2) at relapse to evaluate for changes in CD22 expression pre and post-inotuzumab ozogamicin. Specifically, samples will be evaluated for change in CD22 expression that occurs over time to study the role of CD22 expression as it relates to resistance to therapy or mechanism for relapse. Correlation between changes in CD22 expression and patient's clinical response to inotuzumab ozogamicin as well as cytogenetic/molecular features will be described, in particular to explore the association of CD22-negative subpopulations in patients with KMT2A-rearranged acute lymphoblastic leukemia (ALL).
Change in CD22 site density (Cohorts 1 and 2) | Baseline, post Cycle 1, and at time of relapse
  Exploratory analysis of CD22 will focus primarily on the comparison of paired pre-treatment and post-treatment samples at the following times, 1) End of cycle 1 and 2) at relapse to evaluate for changes in CD22 site density pre and post-inotuzumab ozogamicin. Samples will be evaluated for any change in CD22 site density that occurs over time and to evaluate for the emergence of a CD22 "dim" or "negative" population to study the role of CD22 site density as it relates to resistance to therapy or mechanism for relapse. Correlation between changes in CD22 site density and patient's clinical response to inotuzumab ozogamicin as well as cytogenetic/molecular features will be described, in particular to explore the association of CD22-negative subpopulations in patients with KMT2A-rearranged acute lymphoblastic leukemia (ALL).
Leukemic blast CD22 splice variants (Cohorts 1 and 2) | Baseline, post-Cycle 1, and at time of relapse
  Will be analyzed by ribonucleic acid-sequencing (RNA-Seq). The MAJIQ and VOILA software will be used to identify splicing variations in CD22 from RNA Seq and to quantitate the percent spliced in (PSI) of the alternative exons. CD22 protein levels will be determined by immunoblotting of whole cell protein lysates using several anti-CD22 antibodies recognizing either extracellular or intracellular domains. Both protein sizes and preservation of individual epitopes will be assessed and correlated with alterations in exon inclusion.
Intracellular signaling pathways in leukemic blasts treated with inotuzumab ozogamicin (Cohorts 1 and 2) | Baseline up to 5 years
  Peripheral blood samples will be evaluated by comprehensive protein profiling using CyTOF panels for the two major areas of analyses, surface immunophenotyping to assess the developmental stage of both normal and abnormal B cells and measure their responses to inotuzumab ozogamicin , as well as intracellular epitopes to assess the cellular consequences of treatment with inotuzumab ozogamicin. Exploratory analysis will be performed using Cytobank software tools (viSNE, SPADE and CITRUS) for subpopulations clustering, dimensionality reduction and hierarchical organization.
Changes in peripheral blood absolute B cell numbers and maturation of developing B cell populations with inotuzumab ozogamicin therapy (Cohorts 1 and 2) | Baseline up to 5 years
  Descriptive statistics will be used to characterize patterns of B-cell development including selective loss of subsets. Changes in B cell number and subsets will be described, and exploratory analysis will be conducted to assess their correlation with clinical features including immunoglobulin levels, occurrence of infections, and need for intravenous immunoglobulin (IVIG) replacement during inotuzumab ozogamicin therapy.
Level of MRD by next-generation high-throughput sequencing (HTS) techniques (Cohorts 1 and 2) | Up to 2 cycles
  Compared to MRD measured by flow cytometry. MRD levels at each bone marrow evaluation time point will be measured by standard flow cytometry (MRD-negative defined as < 0.01% or 1 leukemic cell in 10-4 nucleated cells). At the end of cycles 1 and 2, MRD will also be assessed by HTS. The correlation between the measurements with each technique will be described and the sensitivity of flow-based MRD methodology in the setting of CD22-targeted therapy will be explored.
Serum levels of candidate SOS biomarkers Ang2 and L ficolin (Cohorts 1 and 2) | Up to 12 months from last dose of inotuzumab ozogamicin
  Correlated with clinical development of SOS. Descriptive statistics will be used to characterize clinical features of patients experiencing SOS. L-ficolin and Ang2 absolute levels and change in level over time with inotuzumab ozogamicin exposure will be evaluated and correlated with development of SOS. Biomarker levels will be compared using simple comparative statistics between subgroups.
Incidence of SOS in patients who receive prophylaxis with ursodeoxycholic acid (UDCA) during inotuzumab ozogamicin therapy (Cohorts 1 and 2) | Up to 12 months from last dose of inotuzumab ozogamicin
  Descriptive statistics will be used to characterize clinical features of patients experiencing SOS, potential clinical risk factors, and the impact of ursodeoxycholic acid prophylaxis.
Interaction between CAR- T therapy and inotuzumab ozogamicin (Cohorts 1 and 2) | Up to 5 years
  Will be evaluated by incidence of hematologic DLT in patients with CAR-T therapy prior to inotuzumab ozogamicin, incidence of post-inotuzumab ozogamicin CAR-T therapy, time to CAR-T therapy after inotuzumab ozogamicin, and B-cell recovery prior to CAR-T therapy after inotuzumab ozogamicin. Will be summarized using descriptive statistics.
Morphologic response (CR/CRi) (Cohort 2) | Up to 2 cycles (each cycle is 42 days)
  Will be estimated using the proportion of eligible/evaluable patients with CR/CRi response. Analysis will be mostly descriptive.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen M O'Brien, Principal Investigator — Children's Oncology Group
Locations (157):
- United States (156):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Tufts Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

REFERENCES:
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- [Derived] O'Brien MM, Ji L, Shah NN, Rheingold SR, Bhojwani D, Yuan CM, Xu X, Yi JS, Harris AC, Brown PA, Borowitz MJ, Militano O, Kairalla J, Devidas M, Raetz EA, Gore L, Loh ML. Phase II Trial of Inotuzumab Ozogamicin in Children and Adolescents With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia: Children's Oncology Group Protocol AALL1621. J Clin Oncol. 2022 Mar 20;40(9):956-967. doi: 10.1200/JCO.21.01693. Epub 2022 Jan 10. PMID 35007127